CLINICAL TRIAL: NCT02787720
Title: Effects of Varied Rehabilitation Techniques on Survivors of Acute Respiratory Distress Syndrome: A Randomized Controlled Trial
Brief Title: Rehabilitation Techniques on Survivors of Acute Respiratory Distress Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Collaborators: Shahid Beheshti University (Other); Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Vahedian-Azimi, Dr, Baqiyatallah Medical Sciences University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ARDS Rehabilitation
Record Dates: First submitted 2016-05-24; First posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Acute Respiratory Distress Syndrome; Tobacco; Use, Rehabilitation
Keywords: Acute Respiratory Distress Syndrome; Pulmonary Rehabilitation; Rehabilitation Plan; Rehabilitation Techniques; Survivor; Randomized Controlled Trial
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family centered empowerment model (Experimental): The Family-Centered Empowerment Model (FCEM)
  Interventions: Other: Family centered empowerment model
- Continuous care model (Experimental): The Continuous Care Model
  Interventions: Other: Continuous care model

INTERVENTIONS:
Other: Family centered empowerment model — The intervention was conducting Family-Centered Empowerment Model. The intervention package had three steps including pre intervention, during intervention and post intervention. The model has four stages including Perceived threat, Problem solving, Educational partnership, and Evaluation
  Arms: Family centered empowerment model
Other: Continuous care model — The intervention was conducting Family-Centered Empowerment Model. The intervention package had three steps including pre intervention, during intervention and post intervention. The model has four stages including Orientation, Sensitization, Control, and Evaluation
  Arms: Continuous care model

SUMMARY:
A randomized controlled blinded study in patients treated for Acute Respiratory Distress Syndrome (ARDS) in the mixed medical-surgical intensive care units (ICU) of four academic teaching hospitals in Tehran, Iran were conducted to examine the effects of Varied Rehabilitation Techniques on Survivors of ARDS patients. Patients were randomized in the emergency department at the time of ICU admission to one of four groups labeled groups 1, 2, 3 and 4, respectively.

DETAILED DESCRIPTION:
The intervention package had three phases including pre-intervention, intervention, and post-intervention phases. Pre-intervention: During the pre-intervention phase, patients completed the quality-of-life assessment (SF-36), perceived stress questionnaire (PSQ-14), and State and Trait Anxiety, Barthel Index (BI) and Kessler Psychological Distress Scale (K10) questionnaires as well as a Six-minute walk test (6MWT), and 51 times walking per 5 years (at discharge, month 1 to month 42 (each month), and months 45, 48, 51, 54, 57, 60, 63, and 66). A rehabilitation plan was formulated incorporating considerations for the patient's identified strengths' and weaknesses. See the RP section.

Intervention: Once discharged, patients called their study nurse every 2 days to report any problems or complications. Patients were evaluated by their primary multidisciplinary medical team including their pulmonologist, intensivist, internist, psychologist, psychiatrist, physical therapist, and occupational therapist on a weekly basis and at 30 days. At each visit, the patient was interviewed, underwent a physical examination, pulmonary-function testing (PFT), posterior-anterior and lateral (PA-Lat) chest radiography (CXR), resting oximetry, a standardized 6MWT with continuous oximetry, free walking test as long as the stamina and capability of patient, and laboratory tests as indicated. At other times, if patients experienced a problem or complication, they notified investigators and presented to either their multidisciplinary medical team or their primary care provider for evaluation. Patients in the group 1 received rehabilitation employing the mixed model: Family-Centered Empowerment Model (FCEM) and Continuous Care Model (CCM). Group 2 received rehabilitation employing the FCEM, and Group 3 employed CCM, each in 4 stages. Stage 1 of the intervention was awareness and cognition. The patient was evaluated for their insight into their perceived illness severity and perceived sensitivity, or the degree to which they felt threatened by their illness. This was performed by means of 3-5 group sessions in the pre-intervention phase. Group sessions included 3-5 patients and lasted for 45-60 min each. Session content included assessments of the participants' psychological and physical conditions as well as their attitude towards the nature, definition, risk factors, symptoms, medical and nursing care, and complications resulting from the ARDS. In stage 2, patients were assessed for their expectations over 3-5 one-hour sessions. Groups of 3-4 patients shared and learnt from each other under the moderation and guidance of the principal researcher. In stage 3, the degree of patient acceptance was assessed using an educational participation method in group discussion. Patients reached practical solutions through using the problem-solving findings of the previous stage. Stage 4 consisted of formative and summative evaluations. The aim of the formative evaluation was to encourage patients to internalize their locus of control by encouraging personal responsibility about issues of health and seeing his/her self-empowerment. Summative evaluations were performed to evaluate the influence of the intervention on the study's medical outcomes. The study's medical outcomes were assessed in pre intervention, measurement 2 (10-day post intervention), measurement 3 (three-month post measurement 2), and ten following ups includes six three-month periods (6, 9, 12, 15, 18, 21), four six-month periods (27, 33, 39, 45), and two twelve-month period (57, and 69) after intervention by deploying FCEM and CCM questionnaires.

Post-intervention follow-up: Phase 3 began 90 days following pre-intervention (control group), and 90 days after measurement 3 in three intervention groups. To assess the durability and stability of patient empowerment, patient knowledge, attitude and practice (KAP) was assessed over ten follow-up sessions with mentioned intervals. During the 66-month follow-up period, patients attended a total of 56 support-group webinars addressing topics including returning to work, intimate relationships, nutrition, sleep hygiene, tobacco use, exercise, and leisure activities as well as testing and laboratory issues. Follow-up interviews were conducted during home visits, when available, or with the assistance of telephone, Skype, Viber or WhatsApp according to patient preference.

Role of the Designee: Following informed consent, the designated family member or friend (hereafter called designee) continued through the study with the patient as a 'unit'. The designee attended the patient's educational sessions during stages 3 and 4, with stage 2 being according to the family member preference. Recall that stage 2 deals with patient expectations, stage 3 with patient acceptance and problem-solving, and stage 4 with evaluations and internalizing his/her locus of control. The designee and the patient attended the same sessions, and studied the same learning materials. Up to eight family members were allowed to join in the educational sessions if requested. In stage 3, the designee was charged with learning and reinforcing educational material with the patient. In stage 4, when instructed by study investigators, the designee would administer the KAP assessments to the patient. In addition to scores, the designee would provide additional information on the patient's home situation and current condition. Patients were assigned a code, and de-identified data were transmitted from the designee to investigators either by encrypted email, telephone, mail or in person.

Rehabilitation plan: All patients had similar inpatient rehabilitation programs. For patients in the three intervention groups, outpatient rehab included daily exercise for 0-2 h/day. Exercise occurred between 8:00 and 10:00, and types included walking, jogging, bicycle, swimming, or other exercise according to patient preference or resource availability and confirmed by multidisciplinary medical team. Daily exercise was supervised by designated family members. Investigators randomly attended sessions in an unannounced fashion. Although not routinely involved, multidisciplinary medical team consultations were available on investigator request. Exercise data were independently collected from the patient and their designated family member on a weekly basis (κ statistic=0.94). To measure the patients' walking distance, investigators provided them with a Fit bit (Fit bit, San Francisco, USA). Routine care included education on smoking cessation and education on food selection. Patients were provided printed materials, with dietician assessments available on request. Patients in the control group received the same education and printed materials during their inpatient course. Patients exercised daily, at any time, for ≤2 h according to patient tolerance. Sessions were supervised by family members. Investigators did not attend sessions. Exercise data were independently collected from the patient and their designated family member on a weekly basis (κ statistic=0.22). Again, walking distance was measured using the Fit bit. Routine care included education on smoking cessation and education on food selection. Patients were provided printed materials, with dietician assessments available on request.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Informed consent
* Willingness of designated family member or friend to participate
* Has basic health literacy and can fill out questionnaire
* Admitted to the ICU, (6) full code status
* Met ARDS criteria

Exclusion Criteria:

* Patients with any limitation of code status
* Patients who were immobile prior to ICU admission
* Patients who were received prior pulmonary rehabilitation
* Patients who had a documented neurologic or psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-12; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Quality of life: The short form health survey questionnaire with 36 questions | Five years

SECONDARY OUTCOMES:
The 14-Item Perceived Stress Questionnaire | Five years

OTHER OUTCOMES:
The Beck 20-Item state and 20-Item trait anxiety Questionnaires | Five years
the Barthel with 10 variables describing activities of daily living ( ADL) and mobility | Five years
The Kessler Psychological Distress Scale (K10) | Five years
The standardized 6MWT | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Amir Vahedian-azimi, Postdoc, Principal Investigator — Baqiyatallah Universiy of Medical Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rahimi-Bashar F, Salesi M, Gohari-Moghadam K, Jouzdani AF, Pourhoseingholi MA, Vahedian-Azimi A. Assessment of 5-year outcomes of life satisfaction in survivors after rehabilitation programs: a multicenter clinical trial. Sci Rep. 2022 Jan 27;12(1):1497. doi: 10.1038/s41598-022-05355-z. PMID 35087117